CLINICAL TRIAL: NCT05583903
Title: Usability and Acceptability of Virtual Reality-based Cognitive Stimulation by Healthy Participants
Brief Title: Usability, Acceptability, and Safety of Virtual Reality-based Cognitive Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Methodist Hospital Research Institute (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Hina Faisal, Assistant Professor of Clinical Surgery, The Methodist Hospital Research Institute
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: PRO00033195; R03AG078857 (NIH)
Record Dates: First submitted 2022-10-07; First posted 2022-10-18 (Actual); Results first posted 2023-11-21 (Actual); Last update posted 2023-11-21 (Actual); Status verified 2023-11

CONDITIONS: Virtual Reality
Keywords: Young Healthy Volunteers; Elderly Healthy Volunteers; User-Centered Design; Cognitive Exercises

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual Reality Software Usability in Healthy Volunteers Age 18-35 Years (Experimental): Healthy volunteers between the ages of 18 and 35 years will utilize the ReCognition virtual reality software
  Interventions: Other: Virtual Reality Software
- Virtual Reality Software Usability in Healthy Volunteers Age 60 or Greater Years (Experimental): Healthy volunteers 60 years of age and older will utilize the ReCognition virtual reality software
  Interventions: Other: Virtual Reality Software

INTERVENTIONS:
Other: Virtual Reality Software — The ReCognition virtual reality software is delivered via an Oculus Quest 2 device. This three-dimensional simulated software was designed to improve attention and executive functions.
  Other Names: ReCognition Virtual Reality Software

SUMMARY:
This study aims to determine feasibility, acceptability, and usability, and to assess the safety of using a virtual reality-based software called ''ReCognitionVR'' in healthy volunteers.

DETAILED DESCRIPTION:
Virtual reality (VR) imitates reality by creating an artificial 3-D environment using computing technology or software. Using this software with a headset, a virtual environment is created, which cognitively stimulates the user's brain to think they are in an artificial world. Creating a virtual environment allows flexibility and measurement of different types of stimuli while recording the various responses provided by users in the controlled virtual environment. VR strengthens the brain's ability to focus, learn, and retain experience. VR for attention deficit disorders has been reported to have promising results. This trial aims to follow in similar footsteps using the gamification of exercises for cognitive stimulation in healthy volunteers to record outcomes and perform usability testing. These exercise "games" allow users to focus and pay attention to the game while helping reorient and cognitively stimulate the user's brain. The games are built with increasing difficulty and complexity of user demand and output. A novel, 3D-simulated software platform prototype called ''ReCognitionVR'' was developed to provide VR-based cognitive exercises to healthy participants for testing.

The premise of this trial is that VR-based cognitive stimulation software will allow the controlled delivery of structured cognitive exercises focusing on orientation, attention, memory, and executive functions. The system will allow customized frequency and duration of cognitive exercises based on the users' difficulty level in a delightfully relaxed- environment with music.

According to our institutional review board recommendations, this pilot study will be conducted in two steps on two different cohorts which are as follows:

In the first step, the usability, acceptability, and safety of ReCognitionVR-based cognitive exercises will be evaluated on elderly healthy subjects. This study's results will inform the design of a second-step pilot study.

In the second step, the usability, acceptability, and safety of ReCognitionVR-based cognitive exercise will be evaluated for elderly surgical patients who are at high risk for the development of delirium.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-35 years or ≥60 years
* Healthy volunteers who meet one of the following criteria according to their self-reported medical history:

  1. American Society of Anesthesiologists (ASA) 1: A normal healthy patient. Example: Fit, nonobese (BMI under 30), a nonsmoking patient with good exercise tolerance.
  2. ASA 2: A patient with mild systemic disease. Example: Patient with no functional limitations and a well-controlled disease (eg, treated hypertension, obesity with BMI under 35, frequent social drinker, but is nonsmoking).

Exclusion Criteria:

* Age <18 years; 36-59 years
* Person with active psychiatric disorders, especially schizophrenia
* Person who is deaf or blind

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2022-08-14 (Actual); Primary Completion 2023-05-31 (Actual); Study Completion 2023-06-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Houston Methodist Research Institute, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of 30 enrolled participants, 29 met inclusion criteria. One participant in Arm 2 (Virtual Reality Software Usability in Healthy Volunteers Age 60 or Greater Years) completed the study but was outside the limit for BMI and could not be counted in the efficacy endpoints. However, because they completed the study, they were counted in the safety endpoints only.
Groups:
- Virtual Reality Software Usability in Healthy Volunteers Age 18-35 Years (ASA1): Healthy volunteers between the ages of 18 and 35 years will utilize the ReCognition virtual reality software
  Virtual Reality Software: The ReCognition virtual reality software is delivered via an Oculus Quest 2 device. This three-dimensional simulated software was designed to improve attention and executive functions.
- Virtual Reality Software Usability in Healthy Volunteers Age 60 or Greater Years (ASA2): Healthy volunteers 60 years of age and older will utilize the ReCognition virtual reality software
  Virtual Reality Software: The ReCognition virtual reality software is delivered via an Oculus Quest 2 device. This three-dimensional simulated software was designed to improve attention and executive functions.
Period: Overall Study
Arm/Group | Virtual Reality Software Usability in Healthy Volunteers Age 18-35 Years (ASA1) | Virtual Reality Software Usability in Healthy Volunteers Age 60 or Greater Years (ASA2)
Started | 15 | 15
Completed | 15 | 15
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Virtual Reality Software Usability in Healthy Volunteers Age 18-35 Years (ASA1) | Virtual Reality Software Usability in Healthy Volunteers Age 60 or Greater Years (ASA2) | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 28 [25 to 31] | 65 [62 to 67] | 47.5 [28 to 65]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 9 | 13
  Male | 11 | 6 | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 14 | 14 | 28
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 6 | 6 | 12
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 2 | 2
  White | 9 | 5 | 14
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 2 | 2
Body Mass Index, continuous [Median (Inter-Quartile Range); unit: kg/m2] | 23.6 [21.3 to 25.1] | 25.2 [23.8 to 29.3] | 24.5 [22.3 to 26.5]
Non-smoker [Count of Participants; unit: Participants] | 15 | 15 | 30
History of hypertension [Count of Participants; unit: Participants] | 0 | 6 | 6
History of diabetes [Count of Participants; unit: Participants] | 0 | 2 | 2
History of hypercholesterolemia [Count of Participants; unit: Participants] | 0 | 3 | 3

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Using Virtual Reality Software at 20 Minutes After Start
Description: Whether 70% of participants in each group will complete 20 minutes of use of the ReCognition VR-based software (a binary outcome)
Time Frame: 20 minutes after the start of software use
Measure: Count of Participants; unit: Participants
Arm/Group | Virtual Reality Software Usability in Healthy Volunteers Age 18-35 Years | Virtual Reality Software Usability in Healthy Volunteers Age 60 or Greater Years
Number analyzed (Participants) | 15 | 14
Participants | 15 | 14
Statistical Analysis 1: Comparison: Virtual Reality Software Usability in Healthy Volunteers Age 18-35 Years vs Virtual Reality Software Usability in Healthy Volunteers Age 60 or Greater Years; Test type: Superiority; p = 1.00, Fisher Exact

2. Secondary Outcome: Participants With a System Usability Scale Score >35
Description: The proportion of participants with a System Usability Scale score >35 on a scale of 0-100, where higher scores mean better usability.
Time Frame: After completion of use of the virtual reality software, up to 2 hours after the start of software use
Measure: Count of Participants; unit: Participants
Arm/Group | Virtual Reality Software Usability in Healthy Volunteers Age 18-35 Years | Virtual Reality Software Usability in Healthy Volunteers Age 60 or Greater Years
Number analyzed (Participants) | 15 | 14
Participants | 11 | 7
Statistical Analysis 1: Comparison: Virtual Reality Software Usability in Healthy Volunteers Age 18-35 Years vs Virtual Reality Software Usability in Healthy Volunteers Age 60 or Greater Years; Test type: Superiority; p = 0.26, Fisher Exact

3. Secondary Outcome: Participant High Score in Easy Mode
Description: Participant highest score achieved utilizing the virtual reality software, on a scale of 0 to 100, where higher scores indicate better performance in the software game.
Time Frame: After completion of use of the virtual reality software, up to 2 hours after the start of software use
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Virtual Reality Software Usability in Healthy Volunteers Age 18-35 Years | Virtual Reality Software Usability in Healthy Volunteers Age 60 or Greater Years
Number analyzed (Participants) | 15 | 14
score on a scale | 100 [100 to 100] | 100 [100 to 100]
Statistical Analysis 1: Comparison: Virtual Reality Software Usability in Healthy Volunteers Age 18-35 Years vs Virtual Reality Software Usability in Healthy Volunteers Age 60 or Greater Years; Test type: Superiority; p = 0.57, Wilcoxon (Mann-Whitney)

4. Secondary Outcome: Participant High Score in Medium Difficulty Mode
Description: as for outcome 3
Time Frame: After completion of use of the virtual reality software, up to 2 hours after the start of software use
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Virtual Reality Software Usability in Healthy Volunteers Age 18-35 Years | Virtual Reality Software Usability in Healthy Volunteers Age 60 or Greater Years
Number analyzed (Participants) | 15 | 14
score on a scale | 100 [97 to 100] | 99 [96 to 100]
Statistical Analysis 1: Comparison: Virtual Reality Software Usability in Healthy Volunteers Age 18-35 Years vs Virtual Reality Software Usability in Healthy Volunteers Age 60 or Greater Years; Test type: Superiority; p = 0.2, Wilcoxon (Mann-Whitney)

5. Secondary Outcome: Participant High Score in Hard Mode
Description: as for outcome 3
Time Frame: After completion of use of the virtual reality software, up to 2 hours after the start of software use
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Virtual Reality Software Usability in Healthy Volunteers Age 18-35 Years | Virtual Reality Software Usability in Healthy Volunteers Age 60 or Greater Years
Number analyzed (Participants) | 15 | 14
score on a scale | 100 [97 to 100] | 95 [92 to 98]
Statistical Analysis 1: Comparison: Virtual Reality Software Usability in Healthy Volunteers Age 18-35 Years vs Virtual Reality Software Usability in Healthy Volunteers Age 60 or Greater Years; Test type: Superiority; p = 0.001, Wilcoxon (Mann-Whitney)

6. Secondary Outcome: Change From Baseline in Heart Rate After 10 Minutes of Virtual Reality Software Use
Description: Heart rate measured using a vital sign monitor at baseline (immediately prior to software use) and 10 minutes after software use. Change = 10-minute heart rate - baseline heart rate
Time Frame: Baseline and 10 minutes
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Virtual Reality Software Usability in Healthy Volunteers Age 18-35 Years | Virtual Reality Software Usability in Healthy Volunteers Age 60 or Greater Years
Number analyzed (Participants) | 15 | 15
beats per minute | -0.53 (3.46) | 2.2 (7.59)
Statistical Analysis 1: Comparison: Virtual Reality Software Usability in Healthy Volunteers Age 18-35 Years vs Virtual Reality Software Usability in Healthy Volunteers Age 60 or Greater Years; Test type: Superiority; p = 0.21, Wilcoxon (Mann-Whitney)

7. Secondary Outcome: Change From Baseline in Pulse Oximetry Oxygen Saturation After 10 Minutes of Virtual Reality Software Use
Description: Pulse oximetry oxygen saturation measured using a vital sign monitor at baseline (immediately prior to software use) and 10 minutes after software use. Change = 10-minute oxygen saturation - baseline oxygen saturation
Time Frame: Baseline and 10 minutes
Measure: Mean (Standard Deviation); unit: percent oxygen saturation
Arm/Group | Virtual Reality Software Usability in Healthy Volunteers Age 18-35 Years | Virtual Reality Software Usability in Healthy Volunteers Age 60 or Greater Years
Number analyzed (Participants) | 15 | 15
percent oxygen saturation | -.2 (1.01) | -0.07 (0.59)
Statistical Analysis 1: Comparison: Virtual Reality Software Usability in Healthy Volunteers Age 18-35 Years vs Virtual Reality Software Usability in Healthy Volunteers Age 60 or Greater Years; Test type: Superiority; p = 0.66, Wilcoxon (Mann-Whitney)

8. Secondary Outcome: Change From Baseline in Respiratory Rate After 10 Minutes of Virtual Reality Software Use
Description: Respiratory rate at baseline (immediately prior to software use) and 10 minutes after software use. Change = 10-minute respiratory rate - baseline respiratory rate rate
Time Frame: Baseline and 10 minutes
Measure: Mean (Standard Deviation); unit: breaths per minute
Arm/Group | Virtual Reality Software Usability in Healthy Volunteers Age 18-35 Years | Virtual Reality Software Usability in Healthy Volunteers Age 60 or Greater Years
Number analyzed (Participants) | 15 | 15
breaths per minute | 1.2 (2.62) | 0.93 (2.31)
Statistical Analysis 1: Comparison: Virtual Reality Software Usability in Healthy Volunteers Age 18-35 Years vs Virtual Reality Software Usability in Healthy Volunteers Age 60 or Greater Years; Test type: Superiority; p = 0.77, Wilcoxon (Mann-Whitney)

9. Secondary Outcome: Change From Baseline in Systolic Blood Pressure After 10 Minutes of Virtual Reality Software Use
Description: Systolic blood pressure measured using a vital sign monitor at baseline (immediately prior to software use) and 10 minutes after software use. Change = 10-minute blood pressure - baseline blood pressure
Time Frame: Baseline and 10 minutes
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Virtual Reality Software Usability in Healthy Volunteers Age 18-35 Years | Virtual Reality Software Usability in Healthy Volunteers Age 60 or Greater Years
Number analyzed (Participants) | 15 | 15
mm Hg | 1.47 (12.06) | 0.13 (7.00)
Statistical Analysis 1: Comparison: Virtual Reality Software Usability in Healthy Volunteers Age 18-35 Years vs Virtual Reality Software Usability in Healthy Volunteers Age 60 or Greater Years; Test type: Superiority; p = 0.71, Wilcoxon (Mann-Whitney)

10. Secondary Outcome: Change From Baseline in Diastolic Blood Pressure After 10 Minutes of Virtual Reality Software Use
Description: Diastolic blood pressure measured using a vital sign monitor at baseline (immediately prior to software use) and 10 minutes after software use. Change = 10-minute blood pressure - baseline blood pressure
Time Frame: Baseline and 10 minutes
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Virtual Reality Software Usability in Healthy Volunteers Age 18-35 Years | Virtual Reality Software Usability in Healthy Volunteers Age 60 or Greater Years
Number analyzed (Participants) | 15 | 15
mm Hg | -0.33 (5.59) | 1.53 (5.32)
Statistical Analysis 1: Comparison: Virtual Reality Software Usability in Healthy Volunteers Age 18-35 Years vs Virtual Reality Software Usability in Healthy Volunteers Age 60 or Greater Years; Test type: Superiority; p = 0.36, Wilcoxon (Mann-Whitney)

11. Secondary Outcome: Change From Baseline in Heart Rate After Completion of Virtual Reality Software Use
Description: Heart rate measured using a vital sign monitor at baseline (immediately prior to software use) and after completion of the software game. Change = completion heart rate - baseline heart rate
Time Frame: Baseline and the completion of the software game, up to 2 hours
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Virtual Reality Software Usability in Healthy Volunteers Age 18-35 Years | Virtual Reality Software Usability in Healthy Volunteers Age 60 or Greater Years
Number analyzed (Participants) | 15 | 15
beats per minute | -0.4 (3.81) | 1.07 (5.97)
Statistical Analysis 1: Comparison: Virtual Reality Software Usability in Healthy Volunteers Age 18-35 Years vs Virtual Reality Software Usability in Healthy Volunteers Age 60 or Greater Years; Test type: Superiority; p = 0.43, Wilcoxon (Mann-Whitney)

12. Secondary Outcome: Change From Baseline in Pulse Oximetry Oxygen Saturation After Completion of Virtual Reality Software Use
Description: Pulse oximetry oxygen saturation measured using a vital sign monitor at baseline (immediately prior to software use) and after completion of the software game. Change = completion oxygen saturation - baseline oxygen saturation
Time Frame: Baseline and the completion of the software game, up to 2 hours
Measure: Mean (Standard Deviation); unit: percent oxygen saturation
Arm/Group | Virtual Reality Software Usability in Healthy Volunteers Age 18-35 Years | Virtual Reality Software Usability in Healthy Volunteers Age 60 or Greater Years
Number analyzed (Participants) | 15 | 15
percent oxygen saturation | -0.33 (0.82) | 0.00 (0.65)
Statistical Analysis 1: Comparison: Virtual Reality Software Usability in Healthy Volunteers Age 18-35 Years vs Virtual Reality Software Usability in Healthy Volunteers Age 60 or Greater Years; Test type: Superiority; p = 0.23, Wilcoxon (Mann-Whitney)

13. Secondary Outcome: Change From Baseline in Respiratory Rate After Completion of Virtual Reality Software Use
Description: Respiratory rate at baseline (immediately prior to software use) and after completion of the software game. Change = completion respiratory rate - baseline respiratory rate rate
Time Frame: Baseline and the completion of the software game, up to 2 hours
Measure: Mean (Standard Deviation); unit: breaths per minute
Arm/Group | Virtual Reality Software Usability in Healthy Volunteers Age 18-35 Years | Virtual Reality Software Usability in Healthy Volunteers Age 60 or Greater Years
Number analyzed (Participants) | 15 | 15
breaths per minute | 1.07 (2.22) | 0.67 (2.32)
Statistical Analysis 1: Comparison: Virtual Reality Software Usability in Healthy Volunteers Age 18-35 Years vs Virtual Reality Software Usability in Healthy Volunteers Age 60 or Greater Years; Test type: Superiority; p = 0.63, Wilcoxon (Mann-Whitney)

14. Secondary Outcome: Change From Baseline in Systolic Blood Pressure After Completion of Virtual Reality Software Use
Description: Systolic blood pressure measured using a vital sign monitor at baseline (immediately prior to software use) and after completion of the software game. Change = completion blood pressure - baseline blood pressure
Time Frame: Baseline and the completion of the software game, up to 2 hours
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Virtual Reality Software Usability in Healthy Volunteers Age 18-35 Years | Virtual Reality Software Usability in Healthy Volunteers Age 60 or Greater Years
Number analyzed (Participants) | 15 | 15
mm Hg | 5.4 (10.54) | 3.00 (8.07)
Statistical Analysis 1: Comparison: Virtual Reality Software Usability in Healthy Volunteers Age 18-35 Years vs Virtual Reality Software Usability in Healthy Volunteers Age 60 or Greater Years; Test type: Superiority; p = 0.52, Wilcoxon (Mann-Whitney)

15. Secondary Outcome: Change From Baseline in Diastolic Blood Pressure After Completion of Virtual Reality Software Use
Description: Diastolic blood pressure measured using a vital sign monitor at baseline (immediately prior to software use) and after completion of the software game. Change = completion blood pressure - baseline blood pressure
Time Frame: Baseline and the completion of the software game, up to 2 hours
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Virtual Reality Software Usability in Healthy Volunteers Age 18-35 Years | Virtual Reality Software Usability in Healthy Volunteers Age 60 or Greater Years
Number analyzed (Participants) | 15 | 15
mm Hg | -0.07 (6.52) | -3.00 (11.43)
Statistical Analysis 1: Comparison: Virtual Reality Software Usability in Healthy Volunteers Age 18-35 Years vs Virtual Reality Software Usability in Healthy Volunteers Age 60 or Greater Years; Test type: Superiority; p = 0.4, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: The duration of the participant's activity in the study (approximately 20 minutes)
Description: Neurological: Main clusters of cybersickness: gastrointestinal (e.g., stomach awareness, nausea, vomiting), central (e.g., fainting, lightheadedness, blurred vision, disorientation, dizziness), peripheral (e.g., sweating, feeling hot), sopite (e.g., annoyance, drowsiness, tiredness, uneasiness).
  Cardiovascular: New-onset hypotension, bradycardia (HR < 50 bpm), tachycardia (HR >130 bpm)
  Pulmonary: New-onset hypoxia (SpO2 <88%) and tachypnea (respiratory rate >20).
Arm/Group | Virtual Reality Software Usability in Healthy Volunteers Age 18-35 Years | Virtual Reality Software Usability in Healthy Volunteers Age 60 or Greater Years
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 2/15 | 0/15
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Virtual Reality Software Usability in Healthy Volunteers Age 18-35 Years (N=15) | Virtual Reality Software Usability in Healthy Volunteers Age 60 or Greater Years (N=15)
Transient increase in systolic blood pressure (Vascular disorders) | 1 (1) | 0 (0) — Transient >20% increase in systolic blood pressure that did not preclude the participant from completing the study
Transient vague uneasiness (Nervous system disorders) | 1 (1) | 0 (0) — Transient vague uneasiness that did not preclude the participant from completing the study

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-06-05): https://cdn.clinicaltrials.gov/large-docs/03/NCT05583903/Prot_SAP_000.pdf